CLINICAL TRIAL: NCT05978713
Title: A Study to Evaluate Tirzepatide Concentrations in Breastmilk Following Administration of Single Dose of Tirzepatide by Subcutaneous Injection in Healthy Lactating Females
Brief Title: A Study of Tirzepatide (LY3298176) in Healthy Lactating Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18614; I8F-MC-GPIN (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 5 mg Tirzepatide (Experimental): Participants received a single dose of 5 mg tirzepatide injection administered subcutaneously (SC).
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176

SUMMARY:
The main purpose of this study was to look if the study drug, tirzepatide, gets into the breastmilk and, if yes, how long it takes the body to get rid of it from the breastmilk. The study drug was given as a single injection under the skin in healthy lactating females. For each participant, the total duration of the study was approximately 8 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy females as determined by medical evaluation
* Female participants who delivered normal-term infant (at least 37 weeks gestation) and are at least 6 weeks postpartum at the time of screening
* Body mass index (BMI) between 18.5 and 40.0 kilograms per meter squared (kg/m²), inclusive
* Female participants who has well-established lactation and is breastfeeding her infant. Note: Breastfeeding must be discontinued prior to the administration of tirzepatide on Day 1 and not resumed for the remaining duration of the study until a follow-up visit (or for total of 29 days after tirzepatide dosing for participants who discontinue early).

Exclusion Criteria:

* Have a history of inadequate lactation (for multiparous females who have previously breastfed)
* Have confirmed type 1 or type 2 diabetes mellitus
* Regularly use known drugs of abuse or show positive findings on drug screen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 11 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Las Vegas Clinical Research Unit - PPD, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5 mg Tirzepatide
Started | 11
Received a Dose of Tirzepatide | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- 5 mg Tirzepatide: Participants received a single dose of 5 mg tirzepatide injection administered SC.
Arm/Group | 5 mg Tirzepatide
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve of Tirzepatide in Breastmilk From Zero to Infinity (AUC [0-∞])
Description: PK: AUC (0-∞) of Tirzepatide excreted in Breastmilk
Time Frame: Predose, 3, 6, 9, 12, 16, 24, 36, 48, 72, 96, 120, 168, 336, 504, 672 hours post-dose
Population: Participants who received a dose of tirzepatide were eligible for this outcome analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hours per milliliter (ng*h/mL)
Arm/Group | 5 mg Tirzepatide
Number analyzed (Participants) | 11
nanogram*hours per milliliter (ng*h/mL) | NA (NA) — For all participants, insufficient quantifiable concentrations, due to data below the level of detection, were available after the maximum observed drug concentration (Cmax) to calculate the elimination phase parameters for breastmilk. Therefore, AUC(0-∞) in breastmilk was not calculated.

ADVERSE EVENTS:
Time Frame: Baseline to the end of follow-up (up to Day 29)
Description: All enrolled participants who received a dose of Tirzepatide.
Arm/Group | 5 mg Tirzepatide
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 11/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Tirzepatide (N=11)
Abdominal discomfort (Gastrointestinal disorders) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (10)
Vomiting (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 4 (5)
Seasonal allergy (Immune system disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 10 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (5)
Lethargy (Nervous system disorders) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT05978713/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT05978713/SAP_001.pdf